CLINICAL TRIAL: NCT04964232
Title: Intraoperative Body Temperature Measurement Using Infrared Camera: Comparison With Esophageal, and Skin Temperatures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1-2020-0083
Record Dates: First submitted 2021-07-01; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Patients Undergoing General Anesthesia
Keywords: core-temperature; non-contact temperature measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temperature monitoring group (Experimental): The core-temperature is simultaneously measured by esophageal body temperature measurement methods, skin surface body temperature measurement methods, and thermal imaging camera.
  Interventions: Device: Infrared Camera; Device: Esophageal Temperature Probe; Device: Skin temperature probe

INTERVENTIONS:
Device: Infrared Camera — The core-temperature is simultaneously measured by esophageal body temperature measurement methods, skin surface body temperature measurement methods, and thermal imaging camera.
Device: Esophageal Temperature Probe — In patients undergoing general anesthesia, the Esophageal temeperature parameters are measured using an Esophageal probe.
Device: Skin temperature probe — In patients undergoing general anesthesia, the skin spot temeperature parameters are measured using an skin adhesive probe.

SUMMARY:
"A method of monitoring body temperature during surgery is to measure esophageal temperature using a catheter. Although this method is known as a method to accurately measure core temperature, it is not recommended for local anesthesia patients and requires an invasive procedure that can be used to monitor body temperature non-invasive as it may feel uncomfortable during placement and maintenance management. Various methods have been developed to measure body temperature noninvasive, such as in the mouth, armpits, skin surfaces, and aural canals. However, developed methods can also cause discomfort to patients in that they attach sensors to their skin.

In this study, we use the esophageal temperature measurement method, the skin contact temperature measurement method, and the IR contactless temperature measurement method to simultaneously measure body temperature and to compare the accuracy of body temperature measurement according to each method."

ELIGIBILITY:
Inclusion Criteria:

1. An adult who underwent endoscopic/laparotomy Hepatectomy of living donor, Pylorus preserving pancreaticoduodenectomy, Renal allograft, Flexible ureterorenoscopic removal of calculus of upper ureter with regular surgery

Exclusion Criteria:

1. Subjects at risk of bleeding due to esophageal probe, and past cranial, esophageal varicose veins surgery.

Ages: 19 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
The accuracy of core-temperature measurements | Intraoperative period about 1 hour
  The accuracy of core-temperature measurements between infrared camera,esophageal probe and skin probe in patients with general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Jeongmin Kim, Principal Investigator — Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sessler DI, Schroeder M, Merrifield B, Matsukawa T, Cheng C. Optimal duration and temperature of prewarming. Anesthesiology. 1995 Mar;82(3):674-81. doi: 10.1097/00000542-199503000-00009. PMID 7879936
- [Background] Hannenberg AA, Sessler DI. Improving perioperative temperature management. Anesth Analg. 2008 Nov;107(5):1454-7. doi: 10.1213/ane.0b013e318181f6f2. No abstract available. PMID 18931198
- [Background] Wolberg AS, Meng ZH, Monroe DM 3rd, Hoffman M. A systematic evaluation of the effect of temperature on coagulation enzyme activity and platelet function. J Trauma. 2004 Jun;56(6):1221-8. doi: 10.1097/01.ta.0000064328.97941.fc. PMID 15211129
- [Background] Boggan WO, Meyer JS. Effects of serotonergic drugs on methaqualone-induced hypothermia. Res Commun Chem Pathol Pharmacol. 1977 Apr;16(4):629-36. PMID 140451
- [Background] Langesaeter E. Is it more informative to focus on cardiac output than blood pressure during spinal anesthesia for cesarean delivery in women with severe preeclampsia? Anesthesiology. 2008 May;108(5):771-2. doi: 10.1097/ALN.0b013e31816bbe04. No abstract available. PMID 18431110
- [Background] Rajagopalan S, Mascha E, Na J, Sessler DI. The effects of mild perioperative hypothermia on blood loss and transfusion requirement. Anesthesiology. 2008 Jan;108(1):71-7. doi: 10.1097/01.anes.0000296719.73450.52. PMID 18156884
- [Background] Poveda VB, Nascimento AS. Intraoperative body temperature control: esophageal thermometer versus infrared tympanic thermometer. Rev Esc Enferm USP. 2016 Nov-Dec;50(6):946-952. doi: 10.1590/S0080-623420160000700010. English, Portuguese. PMID 28198959
- [Background] Callanan D. Detecting fever in young infants: reliability of perceived, pacifier, and temporal artery temperatures in infants younger than 3 months of age. Pediatr Emerg Care. 2003 Aug;19(4):240-3. doi: 10.1097/01.pec.0000086231.54586.15. PMID 12972820
- [Background] Morley CJ, Hewson PH, Thornton AJ, Cole TJ. Axillary and rectal temperature measurements in infants. Arch Dis Child. 1992 Jan;67(1):122-5. doi: 10.1136/adc.67.1.122. PMID 1739325
- [Background] Muma BK, Treloar DJ, Wurmlinger K, Peterson E, Vitae A. Comparison of rectal, axillary, and tympanic membrane temperatures in infants and young children. Ann Emerg Med. 1991 Jan;20(1):41-4. doi: 10.1016/s0196-0644(05)81116-3. PMID 1984726
- [Background] Cattaneo CG, Frank SM, Hesel TW, El-Rahmany HK, Kim LJ, Tran KM. The accuracy and precision of body temperature monitoring methods during regional and general anesthesia. Anesth Analg. 2000 Apr;90(4):938-45. doi: 10.1097/00000539-200004000-00030. PMID 10735803
- [Background] Jean-Mary MB, Dicanzio J, Shaw J, Bernstein HH. Limited accuracy and reliability of infrared axillary and aural thermometers in a pediatric outpatient population. J Pediatr. 2002 Nov;141(5):671-6. doi: 10.1067/mpd.2002.127664. PMID 12410196
- [Background] Negishi T, Abe S, Matsui T, Liu H, Kurosawa M, Kirimoto T, Sun G. Contactless Vital Signs Measurement System Using RGB-Thermal Image Sensors and Its Clinical Screening Test on Patients with Seasonal Influenza. Sensors (Basel). 2020 Apr 13;20(8):2171. doi: 10.3390/s20082171. PMID 32294973